CLINICAL TRIAL: NCT05535985
Title: A Prospective Randomized Controlled Study of Acupuncture on Postoperative Delirium in Patients With Diabetes Mellitus
Brief Title: Study of Acupuncture on Postoperative Delirium in Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lingling Ding (Other)
Responsible Party: Sponsor-Investigator, Lingling Ding, Professor, Beijing Hospital of Traditional Chinese Medicine
Organization: Beijing Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHOUFA 2022-2-2232
Record Dates: First submitted 2022-09-01; First posted 2022-09-10 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Acupuncture; Postoperative Delirium (POD); Diabetes Mellitus
Keywords: Acupuncture; Postoperative delirium (POD); Diabetes Mellitus; Regional Cerebral Oxygen Saturation (rSO2)
MeSH Terms: conditions — Emergence Delirium; Diabetes Mellitus | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture group (Experimental): In the acupuncture group, acupoints of Baihui, Shenting, Sishencong will be selected for acupuncture stimulation be anesthesia. The needle will be kept for 30 minutes, during which the needle will be performed once every 10 minutes for 10 seconds each time, 4 times in total. The therapist will give the subject verbal cues before and during the needle manipulation.
  Interventions: Device: acupuncture
- placebo acupuncture group (Placebo Comparator): The patients will be treated with consolation needle. Choose treatment of points that near but without going through the acupoints(upper arm deltoid muscle). Use the Park needle (blunt needle, tip obtuse, when acupuncture the feeling is similar to acupuncture needles into the skin, but it retracts instead of piercing the skin) to conduct acupuncture treatment. The retention time and number of needles will be the same as those in the acupuncture group. The therapist will give the subjects verbal cues before and during the acupuncture manipulation, which further reduces the subjects' doubts about the authenticity of acupuncture in the this group. To ensure the implementation of the blinding method, all patients will be treated independently and avoid contacting with each other.
  Interventions: Device: placebo acupuncture
- control group (No Intervention): The patients will undergoing routine anesthesia without acupuncture treatment.

INTERVENTIONS:
Device: acupuncture — treatment of pain or disease by inserting the tips of needles at specific points on the skin
  Arms: acupuncture group
Device: placebo acupuncture — placebo acupuncture
  Arms: placebo acupuncture group

SUMMARY:
1. To evaluate the effectiveness and safety of acupuncture on POD in diabetic patients undergoing surgery, to provide effective prevention and treatment measures of integrated traditional Chinese and western medicine for reducing the incidence of postoperative delirium in high-risk groups, and to provide clinical basis for further promotion of integrated traditional Chinese and western medicine anesthesia in the future.
2. To investigate the relationship between POD and rSO2 in diabetic patients undergoing surgery. To clarify the predictive value of intraoperative rSO2 monitoring on postoperative cognitive function in patients with diabetes, and to explore the effect of acupuncture on cerebral blood flow perfusion in patients with diabetes.

DETAILED DESCRIPTION:
Postoperative delirium (POD) increases the risk of postoperative dementia and mortality. Cognitive decline is common in patients with diabetes mellitus. As an independent risk factor for POD, diabetes significantly increases postoperative dementia and mortality. Our team found that acupuncture can reduce the incidence of POD in elderly patients, increase regional cerebral oxygen saturation (rSO2), and increase cerebral blood flow perfusion in diabetic patients. In this study, a prospective randomized controlled study with placebo acupuncture will be conducted. Diabetic patients undergoing elective surgery will be divided into acupuncture group, placebo acupuncture group and control group. Acupuncture will be used as the intervention method, and the incidence of POD will be the main therapeutic effect evaluation index to explore the efficacy of acupuncture in the prevention and treatment of POD in diabetic patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia in our hospital
* Expected duration of operation >2h
* Ages 18-60
* With type 2 diabetes
* American Society of Anesthesiologists (ASA) grade 2-3 , no severe respiratory, circulation, liver, kidney, coagulation function abnormalities;
* Expected postoperative hospital stay >3 days
* No history of cerebrovascular accident in the past six months
* The informed consent signed

Exclusion Criteria:

* Unable or unwilling to cooperate with cognitive function scale tests
* MMSE score <24
* Refuse acupuncture treatment or have a history of needle sickness
* With skin damage at the acupuncture sites
* Coagulation dysfunction
* Participated in other clinical studies

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | at 8 a.m. the day after surgery
  assess the incidence of postoperative delirium using the 3-minute diagnostic confusion assessment method (3D-CAM)
Incidence of postoperative delirium | at 16 p.m. the day after surgery
  assess the incidence of postoperative delirium using 3D-CAM
Incidence of postoperative delirium | at 8 a.m. the second day after surgery
  assess the incidence of postoperative delirium using 3D-CAM
Incidence of postoperative delirium | at 16 p.m. the second day after surgery
  assess the incidence of postoperative delirium using 3D-CAM
Incidence of postoperative delirium | at 8 a.m. the third day after surgery
  assess the incidence of postoperative delirium using 3D-CAM
Incidence of postoperative delirium | at 16 p.m. the third day after surgery
  assess the incidence of postoperative delirium using 3D-CAM

SECONDARY OUTCOMES:
Regional Saturation of Oxygenation (rSO2) | baseline
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Regional Saturation of Oxygenation (rSO2) | the time when tracheal intubation finished
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Regional Saturation of Oxygenation (rSO2) | the time when the surgery begins
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Regional Saturation of Oxygenation (rSO2) | 1 hour after the beginning of the surgery
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Regional Saturation of Oxygenation (rSO2) | the time when the surgery ends
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Regional Saturation of Oxygenation (rSO2) | Intraoperative
  The brain oxygen saturation monitoring electrode was attached to the forehead, and the baseline level (T0) was recorded after the reading was stable under the condition of air inhalation. rSO2 readings were recorded after induction (T1), at the beginning of surgery (T2), one hour after the beginning of surgery (T3), at the end of surgery (T4), and after extubation (T5). The maximum and minimum values of rSO2 readings during surgery were recorded, and the area under the rSO2 curve was recorded when the rSO2 reading decreased by 13% from baseline for more than 5 minutes.
  rSO2 values of each time point, maximum and minimum values during surgery.
Visual Analogue Score (VAS) | at 8 a.m. and 16 p.m. daily for 3 days after surgery
  Record VAS. VAS is a psychometric response score. Draw a 10 cm horizontal line on the paper. The end of the line is 0, indicating no pain; the other end is 10, indicating severe pain. The middle part shows different levels of pain.
Blood glucose levels | Entering the operating room, the time when the surgery ends
  record blood glucose levels
Expression of reactive oxygen species (ROS), superoxide dismutase (SOD), S100β in serum | Entering the operating room, the time when the surgery ends
  The inflammation level will be assessed.
Expression of peroxisome proliferators-activated receptor-γcoactivator-1α (PGC-1α) | Entering the operating room, the time when the surgery ends
  assess the expression of PGC-1α

OTHER OUTCOMES:
Height | The 1 day before surgery
  Record the height (in meters) of the patient
Weight | The 1 day before surgery
  Record the weight (in kilograms) of the patient
Mini-mental state examination (MMSE) score | The 1 day before surgery
  Scores are measured by the MMSE, with a maximum score of 30, a score between 27 and 30 is considered normal cognitive function, and a score less than 27 is considered cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Lingling Ding, Doctor, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No